CLINICAL TRIAL: NCT04780035
Title: Multicenter Double-blind Placebo-controlled Comparative Randomized Study of the Tolerability, Safety, Immunogenicity and Prophylactic Efficacy of the EpiVacCorona Peptide Antigen-based Vaccine for the Prevention of COVID-19, With the Participation of 3000 Volunteers Aged 18 Years and Above (Phase III-IV)
Brief Title: Study of the Tolerability, Safety, Immunogenicity and Preventive Efficacy of the EpiVacCorona Vaccine for the Prevention of COVID-19
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Federal Budgetary Research Institution State Research Center of Virology and Biotechnology "Vector" (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: COV/pept-03/20
Record Dates: First submitted 2021-02-25; First posted 2021-03-03 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: COVID-19
Keywords: EpiVacCorona vaccine
MeSH Terms: conditions — COVID-19 | interventions — EpiVacCorona vaccine; Sodium Chloride; Solutions; Injections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group "Vaccine" (Experimental): 2,250 volunteers who will be vaccinated with the EpiVacCorona vaccine, twice intramuscularly at a dose of 0.5 ml.
  Interventions: Biological: EpiVacCorona (EpiVacCorona vaccine based on peptide antigens for the prevention of COVID-19)
- "Control Group" (Placebo Comparator): 750 volunteers who will be vaccinated with a placebo, twice intramuscularly at a dose of 0.5 ml.
  Interventions: Other: Placebo (sodium chloride, a 0.9% solution for the preparation of dosage forms for injections)

INTERVENTIONS:
Biological: EpiVacCorona (EpiVacCorona vaccine based on peptide antigens for the prevention of COVID-19) — The EpiVacCorona vaccine is intended to prevent COVID-19. The vaccine relies on chemically synthesized peptide antigens of SARS-CoV-2 proteins conjugated to a carrier protein and adsorbed on an aluminum-containing adjuvant (aluminum hydroxide).
  The vaccine induces the specific immunity against the SARS-CoV-2 coronavirus following two intramuscular injections spaced 21 to 28 days apart.
  The EpiVacCorona vaccine contributes to the development of protective immunity against SARS-CoV-2 coronavirus following two intramuscular administrations given 21 to 28 days apart.
  Arms: Group "Vaccine"
Other: Placebo (sodium chloride, a 0.9% solution for the preparation of dosage forms for injections) — The use of placebo: intramuscularly twice, given 21 to 28 days apart at a dose of 0.5 ml
  Arms: "Control Group"

SUMMARY:
The objective of the clinical study is to evaluate the tolerability, safety, immunogenicity and prophylactic efficacy of the EpiVacCorona vaccine in volunteers aged 18 and above.

The study tasks are to:

* evaluate the safety of the EpiVacCorona vaccine when administered twice intramuscularly;
* evaluate the tolerability of the EpiVacCorona vaccine when administered twice intramuscularly;
* identify any adverse events to the administration of the EpiVacCorona vaccine;
* investigate the humoral immune response following two doses of the EpiVacCorona vaccine;
* investigate the cell-mediated immune response following two doses of the EpiVacCorona vaccine;
* evaluate the prophylactic efficacy of the EpiVacCorona vaccine when administered twice intramuscularly.

DETAILED DESCRIPTION:
The study will screen a maximum of 4,929 volunteers of both sexes aged 18 and above, of which 3,000 volunteers who meet the inclusion criteria and do not have the exclusion criteria will be randomized:

* 2,250 volunteers who will be vaccinated with the EpiVacCorona vaccine, twice intramuscularly at a dose of 0.5 ml;
* 750 volunteers who will be vaccinated with a placebo, twice intramuscularly at a dose of 0.5 ml.

If volunteers drop out of the study, they will not be replaced. All volunteers will be followed up by an investigator physician for 6 months following the first vaccination in order to identify possible late adverse events. In case the volunteer has any late reactions, he/she will be invited to the clinic to correct his/her condition.

ELIGIBILITY:
Inclusion Criteria:

1. Availability of a signed and dated informed consent of the volunteer to participate in a clinical trial, prior to any of the study procedures.
2. Volunteers (men and women) above the age of 18 years with stable indicators of basic vital functions.
3. Ability to attend all scheduled visits and all planned procedures and examinations.
4. Consent of volunteers to use effective contraceptive methods throughout the study, including the observation period for possible post-vaccination reactions.

Exclusion Criteria:

1. History of severe acute respiratory syndrome (SARS) or Middle East respiratory syndrome (MERS) or another coronavirus infection (HCoV-229E, HCOV-OC43, HCoV-NL63, HCoV-HKU1).
2. History of exposure to confirmed or suspected cases of SARS-CoV-2 infection within 1 month prior to randomization.
3. Positive for IgM or IgG to SARS-CoV-2 as detected during screening.
4. Positive PCR test for SARS-CoV-2 as detected during screening.
5. Clinically and laboratory (according to PCR data) confirmed disease caused by SARS-CoV-2 coronavirus, at the moment or in the past.
6. Serious post-vaccination reaction (body temperature above 40 °C , hyperemia or edema greater than 8 cm in diameter) or complication (collapse or shock-like state that developed within 48 hours after vaccination; convulsions, with or without of a febrile state) to a previous vaccination in the past.
7. Aggravated allergic history (anaphylactic shock, Quincke's edema, polymorphic exudative eczema, atopy, history of serum disease, history of hypersensitivity or allergic reactions to the administration of any vaccines, any known allergic reactions to vaccine components, etc.).
8. Hypersensitivity to any component of the product, allergy to vaccine components.
9. History of vaccination with any vaccine within one month prior to randomization.
10. Previous vaccination with rabies vaccines less than 2 months prior to randomization, or planned vaccination with rabies vaccines within 1 month after immunization with the vaccine under study.
11. Pregnancy or breastfeeding.
12. The military.
13. Persons in custody in detention facilities and those serving sentences in correctional facilities.
14. Children under the age of 18.
15. History of any acute respiratory illness less than 3 months prior to randomization.
16. Acute infectious or non-infectious diseases, exacerbation of chronic diseases less than 4 weeks prior to randomization.
17. History of tuberculosis (pulmonary and extrapulmonary), cancer, autoimmune diseases, skin diseases.
18. Long-term use (more than 14 days) of immunosuppressants, systemic glucocorticosteroids or immunomodulatory drugs within 6 months prior to randomization.
19. Use of immunoglobulin drugs or blood products within 3 months prior to randomization.
20. Chronic diseases of the cardiovascular, bronchopulmonary, endocrine systems, gastrointestinal tract, liver, kidneys, blood, disease of the endocrine system in the exacerbation phase or that in the decompensation phase in the past or as detected during laboratory and imaging examination.
21. History of surgery within 6 months prior to randomization.
22. Participation in other clinical trials less than 3 months prior to randomization.
23. Persons with alcohol or drug abuse (medications or narcotics). Use of more than 10 units of alcohol per week (1 unit of alcohol is equivalent to ½ liter of beer, or 200 ml of wine or 50 ml of alcohol) or history of alcoholism, narcomania or drug (medication) abuse.
24. Mental illness or neurasthenia.
25. Positive test for HIV, viral hepatitis B and C, or syphilis.
26. Premenopausal women (last menstrual period ≤ 1 year prior to signing the informed consent) who are not surgically sterile and women who have reproductive potential but do not use or plan to use approved birth control products throughout the study nor they agree to a urine pregnancy test while participating in the study.
27. Serious concomitant diseases or pathological conditions not listed above, which, according to the investigator's opinion, could complicate the assessment of the study results, including any pathological deviations from the age norms and laboratory norms of blood and urine parameters, clinically significant in the investigator's opinion.

And:

1. The investigator's decision to exclude the volunteer for the benefit of the volunteer.
2. False inclusion (violation of inclusion or non-inclusion criteria) or the appearance of non-inclusion criteria during the study.
3. The decision of the investigator or the Sponsor to exclude the volunteer from the study due to a clinically significant deviation from the protocol/violation of the protocol.
4. Any undesirable phenomenon requiring the appointment of drugs not authorized by the protocol of this study.
5. Volunteer's desire to complete the study early for any reason.
6. Volunteer's failure to show up for a scheduled visit without the warning the investigator or loss of communication with the volunteer.
7. Positive urine drug test and / or alcohol breath test during the visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3000 (Actual)
Dates: Start 2020-11-27 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
The proportion of vaccinated volunteers with no laboratory confirmed symptoms caused by SARS-CoV-2, within 6 months post vaccination versus a placebo | within 6 months after the first vaccination
  The proportion of vaccinated volunteers with no laboratory confirmed symptoms caused by SARS-CoV-2, in combination with one or more of the following symptoms: fever or chills; cough; shortness of breath or labored breathing; fatigue; muscle pain; headache; loss of taste or smell; sore throat; a stuffy nose or runny nose; nausea or vomiting; diarrhea, within 6 months post vaccination versus a placebo
The prophylactic efficacy of the vaccine | 9 months after the first vaccination
  The prophylactic efficacy of the vaccine under study is ≥50% compared to a placebo, with the lower limit of the confidence interval of the point estimate for the primary efficacy variable > 30%

SECONDARY OUTCOMES:
The proportion of volunteers with increased levels of the immune response in terms of geometric mean titers of specific antibodies | 21-28 days after the second vaccination
  The proportion of volunteers with increased levels of the immune response in terms of geometric mean titers of specific antibodies in ELISA is more than 4 times greater 21 to 28 days following the second vaccination
The proportion of volunteers with increased levels of the immune response in terms of specific neutralizing antibody titers | 21-28 days after the second vaccination
  The proportion of volunteers with increased levels of the immune response in terms of specific neutralizing antibody titers in ELISA is more than 4 times greater 21 to 28 days following the second vaccination
The frequency of severe cases of COVID-19 following a single / double vaccination | through the whole study, an average of 9 months
  The frequency of severe cases of COVID-19 following a single / double vaccination (including hospitalization, transfer to an intensive care unit, death, etc.)
Duration of disease | through the whole study, an average of 9 months
  Duration of illness in case of COVID-19 disease
The incidence of asymptomatic COVID-19 following a single / double vaccination | through the whole study, an average of 9 months
  The incidence of asymptomatic COVID-19 following a single / double vaccination (to assess the effectiveness of vaccination in preventing SARS-CoV-2 infection)

CONTACTS AND LOCATIONS:
Overall Officials: Rinat A. Maksyutov, PhD, Study Director — Federal Budgetary Research Institution - State Research Center of Virology and Biotechnology "Vector", Federal Service for Surveillance on Consumer Rights Protection and Human Well-being; Nikita V. Lomakin, Principal Investigator — Federal State Budgetary Institution - Central Clinical Hospital with Polyclinic, Administrative Office of the President of the Russian Federation; Vitaly G. Gusarov, Principal Investigator — Federal State Budgetary Institution - N.I. Pirogov National Medical and Surgical Center, Ministry of Health of the Russian Federation; Maria A. Chukina, Principal Investigator — Federal State Budgetary Research Institution - Academician B.V. Petrovsky Russian Research Center for Surgery; Stanislav A. Terpigorev, Principal Investigator — State Budgetary Healthcare Institution of the Moscow region - M.F. Vladimirsky Moscow Regional Research Clinical Institute; Svetlana B. Erofeeva, Principal Investigator — State Budgetary Healthcare Institution of the Moscow region - Krasnogorsk City Hospital # 1; Olga A. Rychkova, Principal Investigator — State Budgetary Educational Institution of Higher Professional Education - Tyumen State Medical University, Ministry of Health of the Russian Federation; Viktoria Y. Delyan, Associate Professor, Principal Investigator — State Autonomous Healthcare Institution - Clinical City Hospital # 7 of Kazan; Vladimir V. Rafalsky, Principal Investigator — Federal State Autonomous Educational Institution of Higher Education - Immanuel Kant Baltic University (short name: FSAEIHE- I. Kant Baltic Federal University)
Locations (8):
- Russia (8):
  - State Budgetary Healthcare Institution of the Moscow region - Krasnogorsk City Hospital # 1 (short name: SBHI MR KCH # 1), Krasnogorsk, Moscow Oblast
  - Federal State Autonomous Educational Institution of Higher Education - Immanuel Kant Baltic University (short name: FSAEIHE- I. Kant Baltic Federal University), Kaliningrad
  - State Autonomous Healthcare Institution - Clinical City Hospital # 7 of Kazan (short name: SAHI CCH # 7), Kazan'
  - Federal State Budgetary Institution - N.I. Pirogov National Medical and Surgical Center, Ministry of Health of the Russian Federation (short name: FSBI - N.I. Pirogov NMSC, Ministry of Health of the Russian Federation), Moscow
  - Federal State Budgetary Research Institution - Academician B.V. Petrovsky Russian Research Center for Surgery (short name: FSBRI - Academician B.V. Petrovsky RRCS), Moscow
  - Research Center: Federal State Budgetary Institution - Central Clinical Hospital with Polyclinic, Administrative Office of the President of the Russian Federation (short name: FSBI Central Clinical Hospital with Polyclinic), Moscow
  - State Budgetary Healthcare Institution of the Moscow region - M.F. Vladimirsky Moscow Regional Research Clinical Institute (short name: M.F. Vladimirsky SBHI MRRCI), Moscow
  - State Budgetary Educational Institution of Higher Professional Education - Tyumen State Medical University, Ministry of Health of the Russian Federation (short name: SBEIHPE - Tyumen State Medical University, Ministry of Health of Russian Federation), Tyumen

IPD SHARING:
Plan to Share IPD: No